CLINICAL TRIAL: NCT04182828
Title: Effect of Intravenous Lidocaine on Immediate Post-operative Pain, Nausea and Vomiting in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Placebo Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Umer Slote, Principal Investigator, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-1558-5378
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Post-operative Pain; Post-operative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Vomiting | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group(PG) (Placebo Comparator): It will be normal saline 0.9%
  Interventions: Drug: Lidocaine
- Lidocaine Group(LG) (Active Comparator): It will be lidocaine 2%
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — both the drugs will be prepared in same volume, color, consistency and appearance
  Other Names: Normal saline 0.9%

SUMMARY:
Lidocaine is a drug that has multiple uses. One of these is that when intravenously administered it is effective in reducing post-operative pain. The aim of this study is to investigate the beneficial effects of intravenous lignocaine on reducing pain, nausea and vomiting after laparoscopic cholecystectomy. Also, by this research, we are aiming to find a suitable alternative analgesic.

DETAILED DESCRIPTION:
After approval of synopsis from College of Physician and Surgeons of Pakistan (CPSP) and Ethical review committee (ERC) of Aga Khan University Karachi, patients fulfilling the inclusion criteria will be enrolled in the study. Written informed consent will be obtained before the surgery. Patients will be randomly allocated by CTU through computer generated block randomization into either lidocaine group (LG) or placebo group (PG).

The clinical trial unit (CTU) will be responsible to prepare the study drug and placebo in the same volume, color, consistency and packaging and treatment allocation would be done by assigning the study drug and placebo numbers. The staff, patient and the anaesthetists will be blind by the drug allocation. Only the CTU will have the list of randomization and their treatment allocation.

All patient will be given general anesthesia as per standard of care. All patients will be pre-medicated with oral midazolam 7.5 mg one hour before operating room. Standard American Society of Anaesthesiologists (ASA) monitoring (NIBP, ECG, and Pulse Oximetry) will be applied. General anesthesia will be induced by Propofol 2 mg/kg, Nalbuphine 0.1mg/kg and Cis-Atracurium 0.2 mg/kg. Isoflurane 1% - 1.5% in a mixture of oxygen and air (50:50) will be used for maintenance of anesthesia. Before tracheal intubation, patients will receive intravenous bolus injection of the study drug in dose of 1.5mg/kg followed by the continuous infusion at the rate of 1.5mg/kg/hr. via standard computerized programmable infusion pump. The infusion will be continued throughout the surgery and will be stopped after extubation. After intubation, patients' minute ventilation will be adjusted to maintain normocapnia (end tidal CO2 35 - 40 mm of Hg). All patients will be given 1gm of intravenous Paracetamol after induction of anaesthesia. Supplemental analgesia, Nalbuphine 1mg, during surgery will be given if the heart rate and systolic blood pressure increases above 20% of respective baseline values and causes other than pain had been ruled out, which would be at the discretion of the primary anaesthetist. Prophylaxis for nausea and vomiting will be given by Dexamethasone 0.1mg/kg at induction of anaesthesia and Ondansetron 0.1mg/kg after the removal of gall bladder. At the end of surgery, residual neuromuscular blockade will be reversed by 0.05mg/kg of neostigmine and 0.5mg of glycopyrolate. The trachea will be extubated once the patient regained consciousness and then transferred to the post anesthesia care unit (PACU).

In the PACU, each patient will be assessed by the primary investigator for pain, nausea and vomiting at 15, 30, and 60 minutes. If the patient's pain will be equal to 4 or more on the numerical rating scale, he/she will be given Nalbuphine 1mg as a rescue analgesic. Likewise, if the patients has complain of nausea or vomiting, equal to or greater than 2 on Bellvile nausea score, he/she will be given Metoclopramide 10mg as rescue antiemetic. The analgesic and anti-emetic requirement in the ward for the first 6 hr. post-operatively will be recorded by the primary investigator.

The time of arrival at PACU will be recorded as "T1". The discharge time from PACU will also be recorded and would be declared as "T2". The time required for the patient to be discharged from the hospital will be recorded as "TD". TD will be the time when surgical team decides that patient can be discharged from the hospital. The difference between the length of stay in the hospital between the two groups will be calculated as total time spent (in HOURS) in the hospital "TT". It will be the sum of time interval between T1 to T2, and T2 to TD.

TT= (T1+T2+TD)

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic cholecystectomy
* All adults aged between 18 to 65 years
* ASA I and II

Exclusion criteria:

* BMI greater than 35kg/m2
* Allergy to local anesthetic agents
* Patient with or history of arrhythmias
* Patients with SGPT greater than 35 IU/L for females and greater than 45 IU/L for males.
* Patients with chronic renal disease and creatinine greater than 1.5mg/dl.
* Chronic use of opioids
* The surgeries which were converted to open procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-11-24 (Estimated); Study Completion 2020-11-24 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain as assessed on numerical rating scale | upto 6 hours
  Immediate pain after laparoscopic cholecystectomy
Post-operative nausea and vomiting as assessed on Bellville nausea score | upto 6 hours
  feeling of nausea and vomiting after laparoscopic cholecystectomy

SECONDARY OUTCOMES:
Discharge time | upto 24 hours
  discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Dr. M. Umer Slote, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No